CLINICAL TRIAL: NCT03111875
Title: Perioperative Hypothermia and Myocardial Injury After Non-cardiac Surgery
Acronym: PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-1017
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Perioperative Care; Surgery--Complications; Hypothermia; Anesthesia; Myocardial Injury
Keywords: Hypothermia; Intraoperative warming; non-cardiac surgery; myocardial injury
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To maintain blinding, the anesthesia record will be sealed in an opaque envelope before patients leave the post-anesthesia care unit. The envelope will be marked "Do not open until [date 35 days after surgery]." Some hospitals will have electronic records; in those cases, we will ask investigators evaluating postoperative outcomes not to access the anesthesia record.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Routine thermal management (Active Comparator): Patients assigned to routine thermal management will not be pre-warmed and ambient intraoperative temperature will be maintained near 20°C per routine. Only transfused blood will be warmed. An Multi-Position Upper Body Warming Blanket forced-air cover will be positioned over an appropriate non-operative site, but will not initially be activated. Should core temperature decrease to 35.5°C, the warmer will be activated as necessary to prevent core temperature from decreasing further.
  Interventions: Device: routine thermal management
- Aggressive thermal management (Experimental): Patients assigned to aggressive warming will be pre-warmed with a full-body Bair Hugger or Bair Paws cover for ≈30 minutes before induction of anesthesia. The warmer will initially be set to "high" which corresponds to ≈43°C. It will be subsequently adjusted to make patients feel warm, but not uncomfortably so. Patients will be aggressively warmed during surgery to a target intraoperative core temperature between 37 and 37.5°C, using an Multi-Position Upper Body and Full Access Underbody Warming Blankets forced-air covers when clinically practical. All intravenous fluids will be warmed to body temperature.
  Interventions: Device: aggressive warming

INTERVENTIONS:
Device: aggressive warming — Patients will be pre-warming 30 minutes before induction of anesthesia and aggressively warmed during surgery to a target intraoperative core temperature between 37 and 37.5°C.
  Arms: Aggressive thermal management
Device: routine thermal management — A forced-air cover will be positioned but will not initially be activated. The warmer will be activated when core temperature decrease to 35.5°C.
  Arms: Routine thermal management

SUMMARY:
We propose to test the hypothesis that aggressive warming reduces the incidence of major cardiovascular complications, compared to routine care. Half of the participants will be randomly assigned to routine care (core temperature ≈35.5°C), while the other half will receive aggressive warming (>37°C core temperature) in a multi-center trial.

DETAILED DESCRIPTION:
Hypothermia increases sympathetic activation, promotes tachycardia, and causes hypertension - all of which may increase the risk of myocardial injury. Moderate perioperative hypothermia is now uncommon, but mild hyperthermia (≈35.5°C) remains common. Whether aggressive warming to a truly normothermic level (≈37°C) improves outcomes remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for major noncardiac surgery expected to last 2-6 hours;
* Having general anesthesia;
* Expected to require at least overnight hospitalization;
* Expected to have >50% of the anterior skin surface available for warming;
* Have at least one of the following risk factors:

  a. Age over 65 years; b. History of peripheral vascular surgery; c. History of coronary artery disease; d. History of stroke or transient ischemic attack; e. Serum creatinine >175 µmal/L (>2.0 mg/dl); f. Diabetes requiring medication; e. Hypertension requiring medication; g. Current smoking.

Exclusion Criteria:

* Have a clinically important coagulopathy in the judgement of the attending anesthesiologist;
* Are septic (clinical diagnosis by the attending anesthesiologist);
* Body mass index exceeding 30 kg/m2;
* End-stage renal disease requiring dialysis;
* Surgeon believes patient to be at particular infection risk.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5056 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States
- China (10):
  - PUMCH, Beijing
  - West China Hospital Sichuan Univeristy, Chengdu
  - Guangdong General Hospital, Guangzhou
  - Chinese University of Hong Kong, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Nanjing Drum Tower Hospital, Nanjing
  - FDSCC (Fudan University Shanghai, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Oriental Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Investigators are welcome to propose collaborative analyses.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication of the main paper.
Access Criteria: Via corresponding author,

REFERENCES:
- [Derived] Song S, Pei L, Chen H, Zhang Y, Sun C, Yi J, Huang Y. Analysis of hospital and payer costs of care: aggressive warming versus routine warming in abdominal major surgery. Front Public Health. 2023 Nov 2;11:1256254. doi: 10.3389/fpubh.2023.1256254. eCollection 2023. PMID 38026375
- [Derived] Sessler DI, Pei L, Li K, Cui S, Chan MTV, Huang Y, Wu J, He X, Bajracharya GR, Rivas E, Lam CKM; PROTECT Investigators. Aggressive intraoperative warming versus routine thermal management during non-cardiac surgery (PROTECT): a multicentre, parallel group, superiority trial. Lancet. 2022 May 7;399(10337):1799-1808. doi: 10.1016/S0140-6736(22)00560-8. Epub 2022 Apr 4. PMID 35390321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 more patients were enrolled due to potential withdrawal.
Pre-assignment Details: 4 more patients than protocol were enrolled due to potential withdrawal. Thus we have a total of 5056 patients enrolled in the actual trial rather than 5052 specified in the protocol.
Period: Overall Study
Arm/Group | Routine Thermal Management | Aggressive Thermal Management
Started | 2529 | 2527
Completed | 2506 | 2507
Not Completed | 23 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Thermal Management | Aggressive Thermal Management | Total
Number analyzed (Participants) | 2506 | 2507 | 5013
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (8) | 67.4 (8) | 67.3 (8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline data were missing in three patients in the aggressive warming group and four patients in the routine thermal management group.
  Participants
    number analyzed (Participants) | 2502 | 2504 | 5006
    Female | 801 | 836 | 1637
    Male | 1701 | 1668 | 3369
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 23.2 (3) | 23.4 (3) | 23.3 (3)
Type of surgery [Count of Participants; unit: Participants]
  Orthopaedic | 49 | 56 | 105
  Laparoscopic | 1301 | 1313 | 2614
  Open abdominal | 613 | 610 | 1223
  Neurosurgical | 89 | 126 | 215
  Urological | 138 | 138 | 276
  Other | 312 | 261 | 573
  Unknown | 4 | 3 | 7
Type of troponin [Count of Participants; unit: Participants]
  Low-sensitivity T | 199 | 200 | 399
  High-sensitivity T | 825 | 823 | 1648
  Low-sensitivity I | 1482 | 1484 | 2966
Timing of surgery [Count of Participants; unit: Participants]
  Elective | 2432 | 2440 | 4872
  Urgent or emergent | 70 | 64 | 134
  Unknown | 4 | 3 | 7
Risk of surgical site infection [Count of Participants; unit: Participants]
  Any infection risk | 1414 | 1421 | 2835
  Colon resection | 392 | 376 | 768
  Rectal resection | 344 | 378 | 722
  Other abdominal surgeries | 407 | 397 | 804
  Contaminated or dirty-infected wound | 438 | 429 | 867
Cardiac risk [Count of Participants; unit: Participants]
  Any cardiac risk | 1791 | 1755 | 3546
  Hypertension requiring treatment | 1201 | 1234 | 2435
  Diabetes requiring medication (oral or insulin) | 466 | 534 | 1000
  End-stage renal failure requiring dialysis | 2 | 2 | 4
  Peripheral vascular disease | 23 | 28 | 51
  Previous myocardial infarction | 46 | 39 | 85
  Smoker | 610 | 558 | 1168
  Congestive heart failure | 18 | 14 | 32
  Chronic obstructive pulmonary disease | 48 | 52 | 100
Medication use [Count of Participants; unit: Participants] — The use of beta blockers, angiotension converting, and etc., is not exclusive for each patient. For example, a patient could use multiple medications thus any use of the following medication is not the sum of all the medication use number below.
  Participants
    Any use of the following (beta blockers, Angiotension converting, Angiotension receptor, or Statin) | 599 | 606 | 1205
    Beta blockers | 199 | 204 | 403
    Angiotension converting enzyme inhibitors | 128 | 143 | 271
    Angiotension receptor blockers | 197 | 211 | 408
    Statin | 313 | 294 | 607

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Composite Outcome Consisted of Myocardial Injury After Non-cardiac Surgery (MINS), Non-fatal Cardiac Arrest, and All-cause Mortality
Description: The primary outcome was a composite of myocardial injury after non-cardiac surgery, non-fatal cardiac arrest, and all-cause mortality within 30 days of surgery. Myocardial injury was diagnosed when available troponin concentrations exceeded generation-specific and type-specific thresholds and were apparently of ischaemic origin (ie, no other obvious cause for artifactual elevation). We used the following thresholds based on available literature at time of adjudication: 1) non-high-sensitivity (fourth-generation) troponin T ≥0.03 ng/ml2; 2) high-sensitivity troponin T ≥65 ng/L; or high-sensitivity troponin T 20-64 ng/L and an increase ≥5 ng/L from baseline3; 3) high-sensitivity troponin I (Abbott assay) is ≥75 ng/L4; 4) high-sensitivity troponin I (Siemens assay) is
  ≥60 ng/L5; or, 5) troponin I (other assays) greater than local 99th percentiles. Myocardial infarction diagnosis required both troponin elevation and at least one diagnostic symptom or sign.
Time Frame: From the end of surgery to 30 days after surgery
Population: 16 patients were missing in Routine thermal management and 10 patients were missing in aggressive thermal management group.
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Thermal Management | Aggressive Thermal Management
Number analyzed (Participants) | 2490 | 2497
Participants | 239 | 246
Statistical Analysis 1: Comparison: Routine Thermal Management vs Aggressive Thermal Management; Test type: Superiority — common effect; p = 0.69, Mixed Models Analysis; Risk Ratio (RR) = 1.04, 95.6% CI 2-sided [0.87 to 1.24]
Statistical Analysis 2: Comparison: Routine Thermal Management vs Aggressive Thermal Management; Test type: Superiority — average relative effect; p = 0.10, Mixed Models Analysis; Risk Ratio (RR) = 0.68, 95.6% CI 2-sided [0.43 to 1.08]

2. Secondary Outcome: Deep or Organ-space Surgical Site Infection
Description: Surgical site infection is defined by US Centers for Disease Control and Prevention criteria. It is consisted of superficial infection, deep infection, and organ-space infection.
  Superficial infection: Infection involves only skin or subcutaneous tissue of the incision.
  Deep infection: Infection appears to be related to the operation and infection involves deep soft tissues (e.g., fascial and muscle layers) of the incision.
  Organ-space infection: Infection involves any part of the anatomy (e.g., organs or spaces), other than the incision, which was opened or manipulated during an operation.
Time Frame: From the end of surgery to 30 days after surgery
Population: 20 patients were missing on this outcome in aggressive thermal management group and 27 patients were missing in routine thermal management group
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Thermal Management | Aggressive Thermal Management
Number analyzed (Participants) | 2479 | 2487
Participants | 157 | 178
Statistical Analysis 1: Comparison: Routine Thermal Management vs Aggressive Thermal Management; Test type: Superiority; p = 0.25, log-binomial models; The relative risk was estimated using a GEE model to adjust for within-patient correlation across components and log link (to estimate relative risk); Risk Ratio (RR) = 1.13, 98.75% CI 2-sided [0.87 to 1.47]

3. Secondary Outcome: Number of Patients Requiring Intraoperative Transfusion
Description: intraoperative transfusion will be yes if this patient received more than 0 unit of red blood cells.
Time Frame: From surgery start to surgery end
Population: 13 patients missing on this outcome from treatment group and 20 patients missing on this outcome from control group
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Thermal Management | Aggressive Thermal Management
Number analyzed (Participants) | 2486 | 2494
Participants | 236 | 254
Statistical Analysis 1: Comparison: Routine Thermal Management vs Aggressive Thermal Management; Test type: Superiority; p = 0.41, log-binomial models; [statistical method as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.07, 98.75% CI 2-sided [0.87 to 1.33]

4. Secondary Outcome: Duration of Hospitalization
Description: The length of hospital stay in days, censored at 30 days
Time Frame: From the day of surgery to the day of discharge, or 30 days after surgery if the patients is still hospitalized
Population: 35 patients were missing on this outcome from treatment group and 41 patients were missing on this outcome from control group
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Routine Thermal Management | Aggressive Thermal Management
Number analyzed (Participants) | 2465 | 2472
days | 8 [6 to 12] | 8 [6 to 12]

5. Secondary Outcome: Readmission
Description: Readmission to a hospital within a month of surgery
Time Frame: From the end of surgery to 30 days after surgery
Population: 59 patients were missing on this outcome from control group and 45 patients were missing on this outcome from treatment group
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Thermal Management | Aggressive Thermal Management
Number analyzed (Participants) | 2447 | 2462
Participants | 135 | 161

ADVERSE EVENTS:
Time Frame: from end of surgery to postoperative 30 days
Description: Adverse events were tabulated as a measure of safety. We considered unexpected safety events that were not predefined outcomes to be adverse events. Events were designated serious when they prolonged hospitalisation or were life threatening. Events were reported by site investigators to the central coordination site at the Cleveland Clinic. Each was independently designated as serious or not by two investigators (EYA, MCC, FA-C, and SML) who were blinded to treatment allocation.
Arm/Group | Routine Thermal Management | Aggressive Thermal Management
All-Cause Mortality (participants affected / at risk) | 24/2506 | 18/2507
Serious Adverse Events (participants affected / at risk) | 30/2506 | 17/2507
Other Adverse Events (participants affected / at risk) | 24/2506 | 22/2507
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Routine Thermal Management (N=2506) | Aggressive Thermal Management (N=2507)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
blood transfusion issue (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — AMET was called during blood transfusion. Temp was noted to be 1 degree high and pt complained of abdominal and back pain and chills, tachy to the 130s. Transfusion was stopped, analgesia provided, and cardiac enzymes were negative.
hypotension (Cardiac disorders) | 6 (6) | 4 (4) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
diarrhea or ilues (Gastrointestinal disorders) | 2 (2) | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Intraoperative liver rupture, abdominal bleeding (Hepatobiliary disorders) | 1 (1) | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
infection (Infections and infestations) | 1 (1) | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Injury (Injury, poisoning and procedural complications) | 10 (10) | 7 (7) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
vascular disorder (Vascular disorders) | 0 (0) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
OTHER ADVERSE EVENTS (reported when occurring in more than 0.003% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Routine Thermal Management (N=2506) | Aggressive Thermal Management (N=2507)
Cardiac disorders (Cardiac disorders) | 5 (5) | 5 (5) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
General disorders (General disorders) | 1 (1) | 3 (3) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Infections and infestations (Infections and infestations) | 1 (1) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 10 (10) | 8 (8) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Vascular disorders (Vascular disorders) | 1 (1) | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03111875/Prot_SAP_000.pdf